CLINICAL TRIAL: NCT04527016
Title: Effects of Airway Microbiota and Blood Eosinophils Based Therapy or Treatment Using Current Clinical Guidelines in Recurrent Preschool Wheeze
Brief Title: Airway Microbiota Based Treatment of Asthma in Preschool Children
Acronym: AMBT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: QYY1.0
Record Dates: First submitted 2020-08-22; First posted 2020-08-26 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Asthma in Children
Keywords: preschool wheeze; airway microbiota
MeSH Terms: interventions — Microbiota

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microbiota and eosinophils phenotype based therapy (Experimental): The children will be treated with different protocol(Fluticasone propionate (FP),Azithromycin,or FP+Azithromycin) according to their Blood eosinophils level and airway microbiota pattern for 3 months and follow up for 1 year.
  Interventions: Procedure: Microbiota and eosinophils based therapy
- Clinical guidelines based therapy (Active Comparator): The children will be treated as directed by their paediatrician, the clinical practice is based on the guideline for the diagnosis and optimal management of asthma in children of China 2016 (FP or montelukast for 3 months，or intermittent budesonide inhalation suspension during wheezing episode) and follow up for 1 year.
  Interventions: Drug: Clinical guidelines based therapy

INTERVENTIONS:
Procedure: Microbiota and eosinophils based therapy — 1. Blood eosinophils ≥3%+ mixed airway microbiota: 3 month course of FP 50 ug twice daily via spacer
  2. Blood eosinophils<3%+ Moraxella species>40% in airway microbiota: Azithromycin 10mg/kg per day for 3 consecutive days a week for 4 weeks;
  3. Blood eosinophils ≥3%+ Moraxella species>40% in airway microbiota: 3 month course of FP 50 ug twice daily via spacer and Azithromycin 10mg/kg per day for 3 consecutive days a week for 4 weeks;
  4. Blood eosinophils<3%+ mixed airway microbiota: intermittent budesonide inhalation suspension (1mg twice daily) and terbutaline inhalation suspension for 7 days during wheeze episode.
  The participants will be followed up for one year after the intervention.
  Arms: Microbiota and eosinophils phenotype based therapy
Drug: Clinical guidelines based therapy — The children will be treated as directed by their paediatrician ( The clinical practice is based on the guideline for the diagnosis and optimal management of asthma in children of China 2016).The treatment protocols include:
  1. regular inhaled FP 50 ug twice daily via spacer for 3 months;
  2. montelukast(4mg od for 3 months)
  3. intermittent budesonide inhalation suspension (1mg twice daily for 7 days during wheeze episode).
  The participants will be followed up for one year after the intervention.
  Arms: Clinical guidelines based therapy

SUMMARY:
Airway microbiota pattern may related the preschool asthma exacerbation. This is a single-center, randomized-controlled trial, the study will compare the management of preschool wheeze determined by airway microbiota phenotype and blood eosinophils level to the management using current clinical guidelines.

DETAILED DESCRIPTION:
In this study, participants will be children aged 1-5 years who have recurrent wheezing and will be allocated to one of two treatment groups, either current clinical care or airway microbiota and blood eosinophils phenotype based management for 3 months.They will be followed up for one year after the intervention. The primary outcome is the frequency of unscheduled healthcare visit for wheezing, the secondary outcome parameters are events of severe wheezing requiring oral or intravenous steroids, events of emergency department visit and hospital admissions, the changes of Test for Respiratory and Asthma Control in Kids (TRACK) score and Paediatric Asthma Caregiver's Quality of Life Questionnaire (PACQLQ) score.

ELIGIBILITY:
Inclusion Criteria:

* physician diagnosed recurrent wheeze（at least 3 episodes of wheezing or at least one course of oral steroids in the last 6 months）

Exclusion Criteria:

* Any congenital heart disease diagnosed by a physician
* Any chronic respiratory condition other than preschool wheeze (bronchopulmonary dysplasia, bronchiolitis obliteran, congenital airway and lung malformations, bronchomalacia, chronic aspiration) diagnosed by a physician
* Received antibiotic last 6 weeks

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
Frequency of unscheduled healthcare visits for wheezing | from baseline to one year follow-up
  the number of visits for wheezing is recorded by the physician

SECONDARY OUTCOMES:
Frequency of severe wheezing requiring oral or intravenous steroids | from baseline to one year follow-up
  the number of courses of an oral prednisolone or intravenous methylprednisolone started for acute wheezing after consultation with a physician, and is recorded by the physician or confirmed by the medical records
Frequency of emergency department visit | from baseline to one year follow-up
  the number of emergency visit is recorded by the physician and confirmed by the medical records
Frequency of hospital admissions | from baseline to one year follow-up
  the number of emergency visit is confirmed by the medical records
The changes of TRACK score | from baseline to one year follow-up
  assessed by questionnaire
The changes of PACQLQ score | from baseline to one year follow-up
  assessed by questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No